CLINICAL TRIAL: NCT01621672
Title: Myeloma Cure Project: Prospective, Randomized Trial of Indefinite Revlimid Maintenance Versus Observation for Currently Event-Free Patients With Multiple Myeloma Who Have Completed 3 Years of VTD/TD or VTD or VRD Maintenance on Total Therapy 3 (TT3) Trials 2003-33 and 2006-66
Brief Title: UARK 2009-09 Myeloma Cure Project: Prospective Trial of Indefinite Revlimid Maintenance Versus Observation for Currently Event-Free Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110468
Record Dates: First submitted 2012-05-31; First posted 2012-06-18 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Myeloma
Keywords: Revlimid; progression free; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Revlimid (Experimental): Revlimid dosing will be in the morning at the same time each day
  Interventions: Drug: Revlimid
- No further treatment (No Intervention): No treatment control.

INTERVENTIONS:
Drug: Revlimid — 10 mg/day in the morning same time each day
  Other Names: Lenalidomide
  Arms: Revlimid

SUMMARY:
The purpose of this study is to determine in a phase II trial, whether further maintenance therapy with Revlimid can extend the duration of progression-free survival and the duration of complete or near complete response compared to no further therapy beyond the TT3 protocol-prescribed 3 years of maintenance with 1 year of VTD plus 2 years with TD, 3 years with VTD (2003-33) or VRD (2006-66).

DETAILED DESCRIPTION:
Determine the associated toxicities in qualitative and quantitative terms using NCI CTCAE(NCI common terminology for adverse events)

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of all races/ethnicities with multiple myeloma previously enrolled on UARK 2003-33 or 2006-66.
* Participant has completed 3 years of maintenance therapy with one of the three study drugs of VTD or VRD and disease status has remained event free (includes patients who prematurely discontinued maintenance therapy as long as 3 years have elapsed since beginning of maintenance).
* All patients must be ages 18 years of age or greater at the time of signing the informed consent form.
* Participant has adequate hematopoietic reserve, defined as platelets > 50,000/μL (in participants with bone marrow hypoplasia, remaining peripheral blood progenitor cells can be infused to boost hematopoietic reserve prior to enrollment).
* Participant has adequate renal function defined as serum creatinine < 3 mg/dL prior to enrolling on study
* Total bilirubin ≤ 1.5 mg/dL prior to enrolling on study
* AST (SGOT) and ALT (SGPT) ≤ 2 x ULN prior to enrolling on study
* Patient must have signed an IRB-approved informed consent and understand the investigational nature of the study.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®
* Pregnant or nursing women may not participate. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within
* 24 hours of prescribing Revlimid® (lenalidomide; prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Revlimid® (lenalidomide).
* FCBP must also agree to ongoing pregnancy testing.
* Lactating females must agree that they will not breastfeed.
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure,
* Pregnancy Testing Guidelines and Acceptable Birth Control Methods † A female of childbearing potential is a sexually mature woman who:

  * has not undergone a hysterectomy or bilateral oophorectomy
  * has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Any condition that the PI believes, laboratory abnormality, or psychiatric illness that would prevent the subject from being enrolled in the research study.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking Revlimid®)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — UAMS Myeloma Institute for Research & Therapy
Locations (1):
- University of Arkansas for Medical Science-MIRT, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Observation: No treatment
Period: Overall Study
Arm/Group | Revlimid | Observation
Started | 25 | 17
Completed | 25 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revlimid | Observation | Total
Number analyzed (Participants) | 25 | 17 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 11 | 6 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 16 | 12 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 17 | 41
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression was defined as any one or more of the following:
  * Serum M protein increase ≥ 25% from baseline (or an increase of ≥ 1 g/dL if serum M protein was ≥ 5 g/dL at baseline), with an absolute increase of ≥ 0.5 g/dL; or
  * Urine M protein increase ≥ 25% from baseline, with an absolute increase of ≥ 200 mg/24 hrs; or
  * If patient had serum M protein < 1 g/dL, urine M protein < 200 mg/24 hrs, and an involved serum free light chain level ≥ 10 mg/dL at baseline: ≥ 25% increase in the difference between involved and uninvolved serum free light chain level, with an absolute increase of ≥ 10 mg/dL; or
  * Bone marrow plasma cell percentage increase ≥ 25% from baseline, with the absolute plasma cell % ≥ 10%; or
  * New bone lesions or soft tissue plasmacytomas, or definite increase in size of existing bone lesions or soft tissue plasmacytomas; or
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to multiple myeloma.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Revlimid | Observation
Number analyzed (Participants) | 25 | 17
percentage of participants | 88 | 71

ADVERSE EVENTS:
Arm/Group | Revlimid | Observation
Serious Adverse Events (participants affected / at risk) | 18/25 | 17/17
Other Adverse Events (participants affected / at risk) | 25/25 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revlimid (N=25) | Observation (N=17)
Grade 3 Allergic reaction/Hypersensitivity (Immune system disorders) | 1 | 0
Grade 4 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Grade 4 Thrombocyopenia (Blood and lymphatic system disorders) | 2 | 2
Grade 4 Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Grade 3 Skin Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Grade 3 Dysphagia (Gastrointestinal disorders) | 1 | 0
Grade 4 Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 4
Grade 3 Gait/ walking (Musculoskeletal and connective tissue disorders) | 2 | 0
Grade 3 CNS Ischemia (Nervous system disorders) | 1 | 0
Grade 3 Mood alteration (Nervous system disorders) | 1 | 0
Grade 3 Sensory/Neuropathy (Nervous system disorders) | 1 | 2
Grade 3 Extremity/limb (General disorders) | 1 | 0
Gade 3 Hypertension (Cardiac disorders) | 0 | 1
Grade 3 SGPT (ALT) increase (Hepatobiliary disorders) | 0 | 1
Grade 3 Skin Infection UNK ANC (Infections and infestations) | 0 | 1
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Grade 3 Apnea (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Revlimid (N=25) | Observation (N=17)
Grade 1 Rhinitis (Immune system disorders) | 2 | 0
Grade 1 Anemia (Blood and lymphatic system disorders) | 8 | 1
Grade 3 Anemia (Blood and lymphatic system disorders) | 2 | 0
Grade 1 Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 0
Grade 2 Leukopenia (Blood and lymphatic system disorders) | 9 | 0
Grade 1 Fatigue (General disorders) | 2 | 1
Grade 2 Hypothyroidism (Endocrine disorders) | 2 | 0
Grade 1 Constipation (Gastrointestinal disorders) | 2 | 0
Grade 1 Diarrhea (Gastrointestinal disorders) | 3 | 0
Grade 2 Diarrhea (Gastrointestinal disorders) | 2 | 0
Grade 1 Alkaline phosphatase increase (Hepatobiliary disorders) | 3 | 2
Grade 1 Bilirubin increase (Hepatobiliary disorders) | 4 | 1
Grade 1 Hypoalbuminemia (Hepatobiliary disorders) | 17 | 8
Grade 2 Hypoalbuminemia (Hepatobiliary disorders) | 2 | 2
Grade 1 SGOT (AST) increase (Hepatobiliary disorders) | 5 | 4
Grade 1 SGPT (ALT) increase (Hepatobiliary disorders) | 6 | 4
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4
Grade 2 Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Grade 1 Hypokalemia (Metabolism and nutrition disorders) | 5 | 7
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Grade 2 Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 3
Grade 1 Sensory/Neuropathy (Nervous system disorders) | 2 | 1
Grade 2 Sensory/Neuropathy (Nervous system disorders) | 5 | 6
Grade 1 Joint (General disorders) | 2 | 0
Grade 2 Upper Back (General disorders) | 2 | 1
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Grade 1 Creatinine increase (Renal and urinary disorders) | 7 | 7
Grade 2 Creatinine increase (Renal and urinary disorders) | 2 | 0
Grade 1 Allergic reaction/Hypersensitivity (Immune system disorders) | 0 | 1
Grade 1 Hearing (monitoring program) (Ear and labyrinth disorders) | 0 | 1
Grade 2 Hearing (w/o monitoring program) (Ear and labyrinth disorders) | 0 | 1
Grade 2 Anemia (Blood and lymphatic system disorders) | 0 | 2
Grade 2 Fatigue (General disorders) | 0 | 2
Grade 1 Constipation (Gastrointestinal disorders) | 0 | 1
Grade 2 Bilirubin increase (Hepatobiliary disorders) | 0 | 3
Grade 2 SGOT (AST) increase (Hepatobiliary disorders) | 0 | 1
Grade 2 Infection , normal ANC lung (Infections and infestations) | 0 | 1
Grade 2 Lung infection UNK ANC (Infections and infestations) | 0 | 1
Grade 1 Bicarbonate decrease (Metabolism and nutrition disorders) | 0 | 3
Grade 2 Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Grade 1 Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3
Grade 1 Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Grade 2 Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Grade 1 Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Grade 2 Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Grade 1 Gait/walking (Musculoskeletal and connective tissue disorders) | 0 | 1
Grade 2 Dry eye (Eye disorders) | 0 | 1
Grade 2 Extremity/limb (General disorders) | 0 | 1
Grade 1 Muscle (General disorders) | 0 | 1
Grade 1 Neuralgia/peripheral (General disorders) | 0 | 2
Grade 1 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Grade 2 Pulmonary/other (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes